CLINICAL TRIAL: NCT04055376
Title: Chronic Treatment of Alzheimer's Disease With Gamma Frequency Stimulation
Brief Title: Daily Light and Sound Stimulation to Improve Brain Functions in Alzheimer's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1903763319
Record Dates: First submitted 2019-08-05; First posted 2019-08-13 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease; Alzheimer Dementia
Keywords: Alzheimer Disease; Cognitive Impairment; Non-invasive Sensory Stimulation; Light and Sound Stimulation; Gamma
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one of two study groups. Subjects in the first group will use the GENUS device with active settings for 6 or 9 months, and subjects in the second group will use the GENUS device with sham settings for 6 or 9 months. At the end of the 6 or 9 month period, all subjects will be given an option to continue the usage of the GENUS device for additional 6 or 9 months. For these additional 6 or 9 months, the device will be set to active settings for all subjects who choose to remain in the study. A 36-month compassionate use extension will be offered at the completion of all of the study visits.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Daily exposure to active stimulation (Experimental): Subjects in this arm will receive daily exposure to active stimulation
  Interventions: Device: GENUS device (Active Settings)
- Daily exposure to control stimulation (Sham Comparator): Subjects in this arm will receive daily exposure to control stimulation
  Interventions: Device: GENUS device (Sham Settings)

INTERVENTIONS:
Device: GENUS device (Active Settings) — Participants in the experimental group will use the GENUS device configured to active settings for 60 minutes daily over 6 or 9 months. After 6 or 9 months, each participant will be given an option to continue the daily usage of the GENUS device configured to active settings for additional 6 or 9 months.
  Note: Due to the COVID-19 pandemic, participants who have not yet reached the 6-month mark will have their 6 month visit postponed to 9 months.
  Other Names: Gamma frequency stimulation; Light and sound stimulation
  Arms: Daily exposure to active stimulation
Device: GENUS device (Sham Settings) — Participants in the control group will use the GENUS device configured to sham settings for 60 minutes daily over 6 or 9 months. After 6 or 9 months, each participant will be given an option to continue the daily usage of the GENUS device configured to active settings for additional 6 or 9 months.
  Note: Due to the COVID-19 pandemic, participants who have not yet reached the 6-month mark will have their 6 month visit postponed to 9 months.
  Other Names: Gamma frequency stimulation; Light and sound stimulation
  Arms: Daily exposure to control stimulation

SUMMARY:
In this trial, the safety and effect of daily exposure to light and sound stimulation on people with mild Alzheimer's Disease (AD) will be studied.

COVID-19 Amendment: Due to the ongoing suspension of all in-person humans subject research across MIT in response to the COVID-19 pandemic, all enrolled participants who have not completed their 6-month visit will have their visit postponed to 9 months with a follow up at 18 months. Subjects who have completed their 6-month visit will still be instructed to continue and return at Month 12 for an evaluation.

OPTIONAL: If the subject would like to come in for an evaluation between Month 9 and 18, we will invite participants to come on Month 12 to complete cognitive testing and EEG.

DETAILED DESCRIPTION:
After screening for eligibility, subjects will be randomized into one of two study groups in a 1:1 ratio. Each subject will use a non-invasive light and sound device, called the GENUS device, at home for 1 hour per day for 6 or 9 months. The GENUS device, which is composed of a panel with light-emitting diode (LED) illumination and speakers for auditory stimulation, delivers light and sound at different frequencies.

Subjects in the first group will use the device with active settings, and subjects in the second group will use the device with sham settings. After 6 or 9 months of the daily usage of the device, all subjects will be given an option to continue the daily usage for additional 6 or 9 months. For these additional 6 or 9 months, the device will be set to active settings for all subjects who choose to remain in the study.

Over the first 6 or 9 months, cognitive, mental health and memory evaluations will be performed at baseline, after 1 month, after 3 months, and after 6 or 9 months of daily usage of the device. Blood draws as well as hearing and vision tests will be performed at baseline and after 6 or 9 months of daily usage of the device. Magnetic resonance imaging (MRI) and electroencephalogram (EEG) will also be performed at baseline, after 3 months, and after 6 or 9 months of daily usage of the device. For subjects who choose to continue the daily usage of the device for additional 6 or 9 months, MRI, EEG as well as cognitive, mental health and memory evaluations will be performed at the end of the 6 or 9 additional months of daily usage. One month after the completion of the daily usage, EEG as well as cognitive, mental health and memory evaluations will be performed (this will be 7 or 10 months after the start of the study for subjects who choose not to continue the daily usage of the device after the initial 6 or 9 months; this will be 13 or 19 months after the start of the study for subjects who choose to continue the daily usage of the device for additional 6 or 9 months after the initial 6 or 9 months).

Participants who complete the study protocol and finish the final study visit at Month 12 or 19 will be offered a long-term extension for a total of 36 months with yearly follow up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 50 - 100.
* Subject must have mild Alzheimer's disease with a Mini Mental State Exam (MMSE) score of 19 -26.
* Subject is willing to sign informed consent document.
* If subject is deemed to not have capacity to sign the informed consent, he/she will need a legally authorized representative to provide surrogate consent.
* Subjects whose primary residence is within 2 hours of Boston
* Able to complete the 1st month of at home stimulation at their primary residence; if subjects plan to spend more than 1 week away from their primary residence during the trial, their inclusion must be assessed by the research team.

Exclusion Criteria:

* Subjects who do not have healthcare.
* Subjects who are being treated with N-methyl-D-aspartate (NMDA) receptor antagonists (eg. Memantine).
* Subjects on medications that lower seizure threshold such as wellbutrin, ciprofloxacin, levofloxacin, etc.
* Subjects with history of seizure or epilepsy within the past 24 months.
* Subjects with clinically significant suicide risk and/or suicide attempt in the past 12 months.
* Subjects with behavioral problems such as aggression/agitation/impulsivity that might interfere with their ability to comply with protocol.
* Active treatment with one or more anti-epileptic agent.
* Subjects who have had a stroke within the past 24 months.
* Subjects diagnosed with migraine headache.
* Active treatment with one or more psychiatric agent (e.g. antidepressants, antipsychotics, etc).
* Subjects who have an active implantable medical device including but not limited to implantable cardioverter defibrillator (ICD), deep brain stimulator (DBS), cardiac pacemaker, and/or sacral nerve stimulator.
* Subjects who have profound hearing or visual impairment.
* Subjects who have a life expectancy of less than 24 months.
* Subjects who are pregnant.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of at-home light and sound stimulation: amount of time of device usage per day | Over 6 or 9 months (or over 12 or 18 months for subjects who choose to continue the daily device usage for 6 or 9 additional months)
  Feasibility of daily at-home light and sound stimulation will be assessed by keeping track of the amount of time the GENUS device is used per day. The device will automatically log the start and end times of the device usage. The log data will be collected and assessed at the interim analysis time points (Month 1, Month 3) and later time points (Month 6 or 9 and Month 12 or 18).
Safety of daily at-home light and sound stimulation: questionnaire | Over 6 or 9 months (or over 12 or 18 months for subjects who choose to continue the daily device usage for 6 or 9 additional months)
  Safety of daily at-home light and sound stimulation will be assessed by using a daily questionnaire that asks for any adverse effects of the stimulation. The daily questionnaires will be collected and assessed at the interim analysis time point (Month 1) and later time points (Month 6 or 9 and Month 12 or 18).

OTHER OUTCOMES:
Change in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) score | Baseline, Month 1, Month 3, Month 6 , and either Month 7 or Month 12 and Month 13. COVID-19 Amendment:Baseline, Month 1, Month 3, Month 9, and either Month 10 or Month 18 and Month 19.
  The Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-cog) is a 11-item neuropsychological test that assesses the severity of cognitive impairment. The items determine the patient's orientation, memory, language, and praxis. Total score of the 11 items ranges from 0 to 70 (lower score indicates lower cognitive impairment).
Change in Mini Mental State Examination (MMSE) score | Baseline, Month 1, Month 3, Month 6, and either Month 7 or Month 12 and Month 13. COVID-19 Amendment:Baseline, Month 1, Month 3, Month 9, and either Month 10 or Month 18 and Month 19.
  The Mini Mental State Examination (MMSE) is an 11-item test that assesses the cognitive aspects of mental function. The items assess orientation, memory, attention, language, and visual construction. Total score of the 11 items ranges from 0 to 30 (lower score indicates greater cognitive impairment).
Change in Montreal Cognitive Assessment (MoCA) Test score | Baseline, Month 1, Month 3, Month 6, and either Month 7 or Month 12 and Month 13. COVID-19 Amendment:Baseline, Month 1, Month 3, Month 9, and either Month 10 or Month 18 and Month 19.
  Montreal Cognitive Assessment (MoCA) Test is a 30-question test that assesses the cognitive aspects of mental function. The questions assess visuospatial/executive function, naming, memory, attention, language, abstraction, delayed recall, and orientation. Total score ranges from 0 to 30 (lower score indicates greater cognitive impairment).
Change in National Alzheimer's Coordinating Center Uniform Data Set Neuropsychological Battery (UDS V3) score | Baseline and Month 6 (and Month 12 for subjects who choose to continue the daily device usage for 6 additional months). COVID-19 Amendment:Baseline and Month 9 (and Month 18 for subjects who continue the daily device usage for 9 additional months.
  The National Alzheimer's Coordinating Center Uniform Data Set Neuropsychological Battery (UDS V3) assesses cognitive performance in dementia and mild cognitive impairment due to Alzheimer's Disease. The battery includes Craft Story 21 Recall (immediate and delayed), Benson Complex Figure Copy (immediate and delayed), Number Span Tests, Category Fluency, Trail Making Test A/B, Multilingual Naming Test (MINT), and the Verbal Fluency: Phonemic Test.
Change in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) | Baseline, Month 1, Month 3, Month 6, and either Month 7 or Month 12 and Month 13. COVID-19 Amendment:Baseline, Month 1, Month 3, Month 9, and either Month 10 or Month 18 and Month 19.
  The Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) evaluates cognitive function and is scored in 6 domains of functioning: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a 5-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). The total score of the CDR-SB is obtained by summing each of the domain box scores, with scores ranging from 0 to 18 (higher score indicates greater cognitive impairment).
Change in Functional Assessment Scale (FAS) | Baseline and Month 6 (and Month 12 for subjects who choose to continue the daily device usage for 6 additional months). COVID-19 Amendment:Baseline and Month 9 (and Month 18 for subjects who continue the daily device usage for 9 additional months.
  The National Alzheimer's Coordinating Center Functional Assessment Scale (FAS) is a 10-item questionnaire that assesses whether subjects had a difficulty or needed help with activities of daily living in the past 4 weeks at the time of assessment.
Change in Geriatric Depression Scale (GDS) | Baseline and Month 6 (and Month 12 for subjects who choose to continue the daily device usage for 6 additional months). COVID-19 Amendment:Baseline and Month 9 (and Month 18 for subjects who continue the daily device usage for 9 additional months.
  The Geriatric Depression Scale (GDS): Short Form is a brief, 15-item questionnaire in which participants are asked to respond by answering "yes" or "no" in reference to how they felt over the past week. For each item, the answer indicating depression is given one point. Total score of the 15 items ranges from 0 to 15, with scores 0 - 4 considered normal, depending on age, education, and complaints; 5-8 indicating mild depression; 9-11 indicating moderate depression; and 12-15 indicating severe depression.
Change in Neuropsychiatric Inventory Questionnaire (NPI-Q) | Baseline and Month 6 (and Month 12 for subjects who choose to continue the daily device usage for 6 additional months). COVID-19 Amendment:Baseline and Month 9 (and Month 18 for subjects who continue the daily device usage for 9 additional months.
  The Neuropsychiatric Inventory Questionnaire (NPI-Q) is a 12-item structured interview with a caregiver to assess behavioral disturbances. Each item consists of a screening question and sub-questions that are rated "no" (not present) or "yes" (present). Each item is then rated for severity on a 3-point scale including 1 (mild), 2 (Moderate) and 3 (Severe).
Change in blood biomarkers for Alzheimer's Disease | Baseline and Month 6. COVID-19 Amendment: Baseline and Month 9.
  Change in blood biomarkers for Alzheimer's Disease, as assessed by measuring levels of amyloid, tau, and neurofilament light chain in the subject's blood sample.
Change in gene expression in peripheral white blood cells: ribonucleic acid (RNA) sequencing | Baseline and Month 6. COVID-19 Amendment: Baseline and Month 9.
  Change in gene expression in peripheral white blood cells, as assessed by profiling the transcriptome of peripheral white blood cells via ribonucleic acid (RNA) sequencing. The peripheral white blood cells will be isolated and collected from the subject's blood sample.
Change in electroencephalography (EEG) signals | Baseline, Month 3, Month 6, and either Month 7 or Month 12 and Month 13. COVID-19 Amendment: Baseline, Month 3, Month 9, and either Month 10 or Month 18 and Month 19.
  Change in brain waves in the Delta, Theta, Alpha, Beta, and Gamma frequency bands, as assessed by analyzing the electroencephalography (EEG) signals recorded from the subject.
Change in functional Magnetic Resonance Imaging (fMRI) signals | Baseline, Month 3, and Month 6 (and Month 12 for subjects who choose to continue the daily device usage for 6 additional months). COVID-19 Amendment:Baseline, Month 3, Month 9 (and Month 18 for subjects who continue the daily device usage for 9 months).
  Change in functional connectivity and structure of the brain, as assessed by analyzing the functional Magnetic Resonance Imaging (fMRI) signals recorded from the subject.
Total sleep time: Actigraph activity monitor | Over 7 months (or over 13 months for subjects continuing the daily device usage for 6 additional months). COVID-19 Amendment: Over 10 months (or over 19 months for subjects continuing the daily device usage for 9 additional months)
  Total sleep time, as assessed by analyzing the sleep data reported by an Actigraph activity monitor. The activity monitor will be attached to a wristband and worn by the subject through the study completion. The data from the activity monitor will be collected and assessed at the interim analysis time point (Month 1, Month 3) and later time points (Month 6 and either Month 7 or Month 12 and Month 13). COVID Amendment: Data will be collected once every 3-4 months via mail past Month 3 visit.
Sleep efficiency: Actigraph activity monitor | Over 7 months (or over 13 months for subjects continuing the daily device usage for 6 additional months). COVID-19 Amendment: Over 10 months (or over 19 months for subjects continuing the daily device usage for 9 additional months)
  Sleep efficiency, as assessed by analyzing the sleep data reported by an Actigraph activity monitor. The activity monitor will be attached to a wristband and worn by the subject through the study completion. The data from the activity monitor will be collected and assessed at the interim analysis time points (Month 1, Month 3) and later time points (Month 6 and either Month 7 or Month 12 and Month 13). COVID Amendment: Data will be collected once every 3-4 months via mail past Month 3 visit.
Physical activity level: Actigraph activity monitor | Over 7 months (or over 13 months for subjects continuing the daily device usage for 6 additional months). COVID-19 Amendment: Over 10 months (or over 19 months for subjects continuing the daily device usage for 9 additional months)
  Physical activity level, as assessed by analyzing the activity level data reported by an Actigraph activity monitor. The activity monitor will be attached to a wristband and worn by the subject through the study completion. The data from the activity monitor will be collected and assessed at the interim analysis time point (Month 1, Month 3) and later time points (Month 6 and either Month 7 or Month 12 and Month 13). COVID Amendment: Data will be collected once every 3-4 months via mail past Month 3 visit.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Huei Tsai, PhD, Principal Investigator — Massachusetts Institute of Technology; Edward S Boyden, PhD, Principal Investigator — Massachusetts Institute of Technology; Emery Brown, MD, PhD, Principal Investigator — Massachusetts Institute of Technology; Diane Chan, MD, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004
- [Background] Martorell AJ, Paulson AL, Suk HJ, Abdurrob F, Drummond GT, Guan W, Young JZ, Kim DN, Kritskiy O, Barker SJ, Mangena V, Prince SM, Brown EN, Chung K, Boyden ES, Singer AC, Tsai LH. Multi-sensory Gamma Stimulation Ameliorates Alzheimer's-Associated Pathology and Improves Cognition. Cell. 2019 Apr 4;177(2):256-271.e22. doi: 10.1016/j.cell.2019.02.014. Epub 2019 Mar 14. PMID 30879788
- [Background] Adaikkan C, Middleton SJ, Marco A, Pao PC, Mathys H, Kim DN, Gao F, Young JZ, Suk HJ, Boyden ES, McHugh TJ, Tsai LH. Gamma Entrainment Binds Higher-Order Brain Regions and Offers Neuroprotection. Neuron. 2019 Jun 5;102(5):929-943.e8. doi: 10.1016/j.neuron.2019.04.011. Epub 2019 May 7. PMID 31076275
- [Derived] Chan D, de Weck G, Jackson BL, Suk HJ, Milman NP, Kitchener E, Avalos VSF, Quay MJ, Aoki K, Ruiz E, Becker A, Zheng M, Philips R, Firenze R, Geigenmuller U, Hammerschlag B, Arnold S, Kivisakk P, Brickhouse M, Touroutoglou A, Brown EN, Boyden ES, Dickerson BC, Klerman EB, Tsai LH. Gamma sensory stimulation in mild Alzheimer's dementia: An open-label extension study. Alzheimers Dement. 2025 Oct;21(10):e70792. doi: 10.1002/alz.70792. PMID 41137616